CLINICAL TRIAL: NCT04139603
Title: Gebeliğe Bağlı Lumbopelvik Ağrıda İki Farklı Kinezyo Bant Uygulamasının Ağrı ve Fonksiyonel Mobilite Üzerine Etkisi
Brief Title: Effects of Two Different Kinesio Taping Applications on Pain and Functional Mobility in Pregnants With Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Zeynep Kamil Women's and Children's Diseases Training and Research Hospital (Unknown)
Responsible Party: Principal Investigator, İlkim Çıtak Karakaya, PT. PhD. Prof., Prof., Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 47921137-050.01.04-E.109998
Record Dates: First submitted 2019-10-22; First posted 2019-10-25 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Lumbopelvic Pain
Keywords: kinesio tape; pain; functional mobility; ergonomic education; pelvic girdle questionnaire; five times sit to stand test; timed up and go test; stair climb test
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lumbopelvic kinesio taping (LPKT) (Active Comparator): Two I-shaped kinesio tapes in 40 cm length will be applied bilaterally, beginning from 5 cm below the spina iliaca posterior superiors (SIPSs) to the level of the 12th costae, in maximum trunk flexion position, on the paravertebral muscles, by inhibition technique of muscle correction techniques. The tapes will be placed with no tension at 5 cm of both ends, and with 15-25% tension in between. In addition, an extra I-shaped tape will be placed perpendicullar to these tapes with the ligament correction technique, while the pregnant women are in the vertical upright position, at the level of the sacroiliac joints, starting with a tensile strength of 75-100% from the middle, and then with no tension at two ends.
  Interventions: Other: Lumbopelvic kinesio taping
- Abdominal supported lumbopelvic kinesio taping (ALPKT) (Experimental): An abdominal support tape will be added to the LPKT. In order to reduce the tension of the uterus ligaments, and to help perception of the normal elasticity of the target tissues, ligament technique will be used. The middle part of an I-shaped tape will be placed to the midpoint of the lower abdomen, and then will be progressed laterally and above with 50% tension.
  Interventions: Other: Abdominal supported lumbopelvic kinesio taping
- Placebo taping (Placebo Comparator): A Micropore™ surgical plaster of the same color with KT will be applied with no tension, as described in the LPKT technique.
  Interventions: Other: Placebo tapng

INTERVENTIONS:
Other: Lumbopelvic kinesio taping — Kinesio tapes applied to the lumbopelvic region will stay 3 days. They will be removed from the site, and the skin will be checked and cleaned, and then reapplied for the next 3 days.
  An ergonomic education program will be given after the baseline measurements, and will last for 45-60 minutes. A brochure including ergonomic principles with images will also be provided.
  Other Names: Ergonomic education
  Arms: Lumbopelvic kinesio taping (LPKT)
Other: Abdominal supported lumbopelvic kinesio taping — Kinesio tapes applied to the lumbopelvic region and abdominal area will stay 3 days. They will be removed from the sites, and the skin will be checked and cleaned, and then reapplied for the next 3 days.
  An ergonomic education program will be given after the baseline measurements, and will last for 45-60 minutes. A brochure including ergonomic principles with images will also be provided.
  Other Names: Ergonomic education
  Arms: Abdominal supported lumbopelvic kinesio taping (ALPKT)
Other: Placebo tapng — Placebo tapes (just like Kinesio tapes) applied to the lumbopelvic region without any tension will stay 3 days. They will be removed from the site, and the skin will be checked and cleaned, and then reapplied for the next 3 days.
  An ergonomic education program will be given after the baseline measurements, and will last for 45-60 minutes. A brochure including ergonomic principles with images will also be provided.
  Other Names: Ergonomic education
  Arms: Placebo taping

SUMMARY:
This study evaluates and compares the effects of two different kinesio taping applications on pain and functional mobility in pregnancy related lumbopelvic pain.

DETAILED DESCRIPTION:
Literature studies on the effectiveness of kinesio taping (KT) in pregnancy related lumbopelvic pain (LPP) are limited in number and have methodological shortcomings such as lack of randomization, a control group or assessor and/or patient blindness. Although generally presenting a significant effectiveness of KT on intensity of pain and disability, these parameters are evaluated by subjective methods, and the findings do not rely on quantitative data, in general.

In addition, the intervention parameters used in these studies, such as the KT techniques used, amount of KT tension and duration of the intervention are different from each other, and there is lack of studies comparing the effectiveness of different KT techniques.

In this study, effectiveness of two different KT applications will be compared with placebo KT:

1. Lumbopelvic KT (LPKT): Two I-shaped kinesio tapes in 40 cm length will be applied bilaterally, beginning from 5 cm below the spina iliaca posterior superiors (SIPSs) to the level of the 12th costae, in maximum trunk flexion position, on the paravertebral muscles, by inhibition technique of muscle correction techniques. The tapes will be placed with no tension at 5 cm of both ends, and with 15-25% tension in between. In addition, an extra I-shaped tape will be placed perpendicullar to these tapes with the ligament correction technique, while the pregnant women are in the vertical upright position, at the level of the sacroiliac joints, starting with a tensile strength of 75-100% from the middle, and then with no tension at two ends.
2. Abdominal supported LPKT (ALPKT): An abdominal support tape will be added to the LPKT. In order to reduce the tension of the uterus ligaments, and to help perception of the normal elasticity of the target tissues, ligament technique will be used. The middle part of an I-shaped tape will be placed to the midpoint of the lower abdomen, and then will be progressed laterally and above with 50% tension.

For placebo application, a Micropore™ surgical plaster of the same color with KT will be applied with no tension, as described in the LPKT technique.

All participants will undergo a 45-60 minutes of standard ergonomic education after initial assessments and following the first taping applications, They will be observed in regard to their behaviours during different activities such as standing, sitting, walking, turning in bed and standing from the bed. Necessary warnings will be given about correcting their posture and behaviors in terms of ergonomic principles.

ELIGIBILITY:
Inclusion Criteria:

* being able to read and write in Turkish,
* being in 2nd or 3rd trimester of pregnancy,
* having lumbar or pelvic girdle pain for at least one week
* signing the informed consent form for the study

Exclusion Criteria:

* visual, auditory or cognitive problems which may prevent participation to the study
* health problems other than pregnancy related lumbopelvic pain (orthopedic, neurologic, cardiorespiratory, etc.) or trauma history, which may affect standing from sitting, walking or stair climbing activities
* Any gynecological or urological problems which may mimic pregnancy related lumbopelvic pain
* Any ddiagnosed pregnancy complications (preeclampsy, pregnancy related hypertension, diabetes, fetal anomaly, etc.)
* Multiple gestation
* History of spinal injury, ankylosing spondilitis, rheumatoid arthritis, intervertebral disc pathology
* Positive straight leg raising test result or peripheral sensory or motor impairments which may indicate lumbar interbertebral disc pathology
* History of prepregnancy low back pain
* Using any analgesic or myorelaxant medication
* Contraindications to KT (impaired skin integrity or lesion in the lumbopelvic and abdominal regions, history of allergic reaction, etc.)
* previous KT experience

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity during resting | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  0 (no pain)-10 cm (unbearable pain) visual analogue scale will be used.
Change in pain intensity during timed up and go (TUG) test | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  0 (no pain)-10 cm (unbearable pain) visual analogue scales will be used.
Change in pain intensity during five times sit to stand test | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  0 (no pain)-10 cm (unbearable pain) visual analogue scales will be used.
Change in pain intensity during stair climbing test | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  0 (no pain)-10 cm (unbearable pain) visual analogue scales will be used.
Change in time of completing timed up and go test (seconds) | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  All participants will perform the test from a chair (height: 46 cm) with back-support. They will be asked to stand up, walk three meters, turn around, walk back to the chair, and sit down as fast as they can. Time to complete the test will be recorded (sec). Lower times indicate better functional mobility level for walking.
Change in time of completing five times sit to stand test (seconds) | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  The participants will sit on a straight back chair (43 cm height) with arms folded across their chest. They will be instructed to stand up and sit down as quickly as possible 5 times, keeping their arms folded across their chest. Time for completing the test will be recorded (sec). Lower times indicate better functional mobility level for sit to stand activity.
Change in time of completing stair climbing test (seconds) | baseline, approximately one-hour after the first taping, three days after the first taping, and one week after the first taping
  The participants will be asked to ascend and descend 10 stairs. Time of completing the test will be recorded in seconds. Lower times indicate better functional mobility level in stair activities

SECONDARY OUTCOMES:
Change in activity limitation | baseline, three days after the first taping, and one week after the first taping
  Turkish version of Pelvic Girdle Questionnaire will be used. Total score of the questionnaire varies between 0 and 75, and higher scores indicate higher activity limitation.

CONTACTS AND LOCATIONS:
Overall Officials: İlkim Çıtak Karakaya, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Zeynep Kamil Women's and Children's Disease Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reyhan AC, Dereli EE, Colak TK. Low back pain during pregnancy and Kinesio tape application. J Back Musculoskelet Rehabil. 2017;30(3):609-613. doi: 10.3233/BMR-160584. PMID 28035911
- [Background] Kalinowski P, Krawulska A. Kinesio Taping vs. Placebo in Reducing Pregnancy-Related Low Back Pain: A Cross-Over Study. Med Sci Monit. 2017 Dec 26;23:6114-6120. doi: 10.12659/msm.904766. PMID 29277836
- [Background] Kuciel N, Sutkowska E, Cienska A, Markowska D, Wrzosek Z. Impact of Kinesio Taping application on pregnant women suffering from pregnancy-related pelvic girdle pain - preliminary study. Ginekol Pol. 2017;88(11):620-625. doi: 10.5603/GP.a2017.0111. PMID 29303216